CLINICAL TRIAL: NCT06626321
Title: BE IMMUNE: Behavioral Economics to IMprove and Motivate Vaccination Using Nudges Through the EHR, A Replication Trial
Brief Title: Behavioral Economics to Improve Flu Vaccination Using EHR Nudges Replication
Acronym: BE IMMUNE Rep
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Shivan J Mehta, Associate Chief Innovation Officer, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 856739; R33AG068945 (NIH)
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Behavior, Health; Flu; Flu Vaccination
Keywords: Flu Vaccine Uptake; EHR Nudge; Behavioral Economics; Health Disparities
MeSH Terms: conditions — Health Behavior; Influenza, Human

STUDY DESIGN:
Intervention Model Description: We will randomize clinics 2:1 to the nudge arm or control arm using covariate-constrained randomization. Within the high-risk patient subgroups, stratifying by intervention clinics, patients will be randomized 1:1 in Way to Health using permuted block randomization using random block sizes of 2, 4, and 6 to receive the additional intensification bidirectional text messaging nudge or standard messaging.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Clinics randomized to the control arm will receive standard of care.
- Intervention Arm (Experimental): Clinics randomized to the intervention arm will receive the toolkit of clinician and patient facing nudges. Patient nudges will be pre-visit text message reminders (standard messaging content). Clinician nudges will be monthly peer comparison feedback and default pended orders.
  Interventions: Behavioral: Pre-visit patient text messaging; Behavioral: Default pended order; Behavioral: Monthly peer comparison feedback
- High Risk Intensification Arm (Experimental): Patients in the intervention clinics identified as high risk for noncompletion of the flu vaccine will be randomized 1:1 to receive the high risk intensification arm or remain in the standard intervention arm. Patients in the high risk intensification arm will receive an additional bidirectional texting component.
  Interventions: Behavioral: Pre-visit patient text messaging; Behavioral: Default pended order; Behavioral: Monthly peer comparison feedback; Behavioral: High risk bidirectional pre-visit text messaging

INTERVENTIONS:
Behavioral: Pre-visit patient text messaging — Patients will be sent text message reminders 3 days and 24 hours prior to their scheduled primary care visit. The messages will inform the patient that a flu shot has been reserved for them at their upcoming visit and encourage the patient to ask their provider about receiving the vaccine.
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: Default pended order — A default pended order for the flu vaccine will be pended to the patients upcoming primary care encounter and will be visible to the provider during the visit encounter. Clinical staff will have the option of signing the order or dismissing it if they deem it inappropriate for a given patient.
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: Monthly peer comparison feedback — Each month, clinicians will be sent an email containing what percent of their eligible patients received the flu vaccine and how that compares to other peer clinicians in the intervention
  Arms: High Risk Intensification Arm; Intervention Arm
Behavioral: High risk bidirectional pre-visit text messaging — High risk patients randomized to receive the high risk intensification nudge will receive a bidirectional text messaging component prior to their visit. This intervention will query the patient about common questions or concerns about receiving the flu vaccine. If the patient responds, it will provide additional educational materials based on the patient's specific concern(s).
  Arms: High Risk Intensification Arm

SUMMARY:
This study will be a 6-month, cluster randomized, pragmatic replication trial to evaluate the effectiveness of personalized nudges to clinicians and patients, relative to a control, to increase flu vaccination rates among older adults in accordance with CDC guidelines. This will include clinician and patient level nudge interventions, with additional, intensified nudge interventions for patients identified as high risk for not receiving a flu vaccine. Among the intervention clinics, patients will receive pre-visit text message reminders about the flu vaccine, and clinicians will receive a default pended order in the visit encounter in the EHR, along with monthly peer comparison feedback about their flu vaccine completion rate. Patients identified as high risk for noncompletion will be individually randomized to receive an additional bidirectional text message nudge or the standard text messaging

DETAILED DESCRIPTION:
Many older adults are at risk of illness, hospitalization, and death from vaccine-preventable diseases. More than half of older adults in the United States are not vaccinated for flu which has remained relatively constant over the past decade, and there are racial, ethnic, and socioeconomic disparities in care. In this study, we will evaluate personalized nudges to clinicians and patients to help increase flu vaccination rates during primary care visits among older adults at three distinct health systems, with a particular focus on population subgroups at high risk for vaccine noncompletion. In a partnership between Penn Medicine and University of Washington (UW) Medicine, a 6-month, multisite, cluster randomized, pragmatic trial with an additional intensification arm for high-risk patients was conducted from September 2023-February 2024. We will now conduct a 6-month replication trial at Lancaster General Health for the 2024-2025 flu season.

ELIGIBILITY:
Inclusion Criteria:

All patients must meet the following criteria to be eligible:

1. Age ≥ 50 years
2. A scheduled new or return (non-urgent/sick) primary care appointment at one of the study practices at Lancaster General Health
3. Have not received their annual flu vaccine during the active intervention period (September- February)
4. Eligible to receive the flu vaccine

For the patient intensification nudge, at least one of the following criteria must be met to be considered high risk and randomized to receive the intensification nudge:

1. Age ≥ 70 years
2. Living in a lower income community (lowest quartile, zip-code based)
3. Did not receive a flu vaccine in the previous calendar year
4. Self-identifies as Non-Hispanic Black

Clinicians must meet the following criteria to be eligible to receive peer comparison feedback:

1. Practicing physician (MD, DO) or advanced practice provider (NP, PA) with the exception of residents and fellows
2. Have a minimum patient panel of at least 50 patients, and
3. Practicing at a clinical site randomized to receive the clinic-level nudge interventions.

Exclusion Criteria:

Patients will be excluded from the study if they:

1. Have a documented allergy to flu vaccine
2. Have a flu vaccine exclusion modifier in Health Maintenance
3. Have opted out of research according to individual site guidelines and policies
4. Have no phone number (home or mobile) listed in their chart

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26248 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-05-28 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who receive the flu vaccine at the visit | 4 days from enrollment, at the eligible visit
  The primary outcome is flu vaccination completion during the first eligible primary care visit.

SECONDARY OUTCOMES:
Proportion of patients who receive the flu vaccine within 3 months after the visit | 3 months
  The secondary outcome is flu vaccination completion within 3 months after the first eligible primary care visit.

CONTACTS AND LOCATIONS:
Overall Officials: Shivan Mehta, MD, MBA, MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- Lancaster General Health, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share our analytical code(s).
Supporting Information: Study Protocol, Analytic Code
Time Frame: Within one year of trial completion.